CLINICAL TRIAL: NCT03828708
Title: Different Iron Exposure on the Development of Gut Microbiota From Birth to Four Months
Brief Title: Early Iron Exposure on the Gut Microbiota in Young Infants
Acronym: IF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-1317
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Infant Development
MeSH Terms: interventions — Iron; Infant Formula

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the two groups with different amount of iron consumed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard iron arm (Experimental): Participants randomized to this arm will consume infant formula containing 12 mg/L of iron, equivalent to the standard iron content in U.S. infant formula
  Interventions: Other: Iron in infant formula
- Low iron arm (Experimental): Participants randomized to this arm will consume infant formula containing 5 mg/L of iron, equivalent to the standard iron content in European infant formula
  Interventions: Other: Iron in infant formula

INTERVENTIONS:
Other: Iron in infant formula — Participants will receive the same low-iron (5 mg/L) infant formula. Infants in the standard iron group will add iron supplement to pre-made infant formula so the iron content will be 12 mg/L.

SUMMARY:
This study will look at the amount of iron in infant formula and how that affects a child's gut development. The children of mothers who plan to formula feed their children will be randomized to receive either high iron or low iron formula from birth until 4 months of age. Infants will consume only the study provided formula during enrollment. Blood and stool samples will be collected at birth and end of study to measure the effects of the iron exposure. The overall object is to compare high iron versus low iron exposure in formula-fed infants during the first months of life. Aims include determining the types of bacteria that are present in the infants' fecal microbiome, determining the effect of high iron exposure on gut microbiome and sleep patterns, and comparing iron status and homeostasis between the low and high iron formula groups.

DETAILED DESCRIPTION:
Disturbance of the gut microbial colonization during infancy may result in long-term programming impact of metabolism and disease risks of the host. The early gut microbial colonization coincides with the maturation of the infant's mucosal innate immune system and research showed that the gut microbial dysbiosis is associated with impaired innate immune development. Thus, ensuring proper microbial colonization early in life is critical to the maturation of the immune system and long-term health.

Iron fortification can increase the abundance of pathogenic bacteria and induce inflammation in older infants. However, it is still not known what the effect of iron is on a more vulnerable population: the newborn infant, who has immature immune system. Infants 0-4 months are at a low risk for iron deficiency due to the iron endowment at birth, which is compatible with the very low iron content (<0.5mg Fe/L) in breastmilk. However, commercial infant formulas are all fortified with ≥12mg Fe/L. Whether this striking difference drives adverse health effects is unknown/unexamined, especially on early colonization and immune homeostasis. The overall objective is to determine the impact of high vs. low iron exposure in formula-fed infants during the early post-natal months on gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy new born infants

Exclusion Criteria:

* Newborn infants with conditions that prohibit cow-milk based formula consumption

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | birth to 4 months of age
  the gut microbial structure of the participants, by stool samples collected

SECONDARY OUTCOMES:
Iron status: soluble transferrin receptor | at baseline (birth) and end of intervention (4 months)
  Soluble transferrin receptors are proteins found in blood that can be elevated with iron deficiency.
Iron status: ferritin | at baseline (birth) and end of intervention (4 months)
  A ferritin blood test shows how much iron is stored in your body.
Iron status: hepcidin | at baseline (birth) and end of intervention (4 months)
  Hepcidin is a regulator of iron metabolism.
Inflammation: c-reactive protein | at baseline (birth) and end of intervention (4 months)
  C-reactive protein (CRP) is a substance produced by the liver in response to inflammation.
Immunity: soluble CD14 | at baseline (birth) and end of intervention (4 months)
  biomarker of innate immunity
Sleep patterns: duration | end of intervention (4 months)
  Participants will wear a device (Micro Motionlogger Watch version 734) to provide objective measurements of duration.

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Tang, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
the gut microbiome sequencing data will be shared